CLINICAL TRIAL: NCT01860508
Title: Advanced Metastatic Non-small Cell Lung Cancer Patients Aged or PS Score 2 Points for First Line Application Pemetrexed/Carboplatin Chemotherapy Regimens Sequential Pemetrexed Single Drug Maintenance Treatment of Clinical Research and Related Predictive Biomarkers of Exploratory Research
Brief Title: A Study of PC Sequential Pemetrexed Single Drug Maintenance Treatment for NSCLC and Related Predictive Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Attending doctor of medical oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-PEM-WJL
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Progression free Survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pemetrexed (Experimental)
  Interventions: Drug: pemetrexed /carboplatin

INTERVENTIONS:
Drug: pemetrexed /carboplatin

SUMMARY:
PFS

ELIGIBILITY:
Inclusion Criteria:

.≥65 years or PS 2

* Patients who were diagnosed by the histologic, cytologic diagnosis of IV non-small cell lung cancer
* Patients received no chemical therapy or only received targeted therapy,and there is evidence show the patent is PD
* Presence of at least one index lesion measurable by CT scan or MRI

  * leucocyte ≥ 3.5×109/L
  * neutrophil ≥ 1.5×109/L
  * platelet ≥ 80×109/L
  * Hemoglobin ≥ 9g/L
  * ALT and AST ≤ 2.5×ULN ,Tbil≤ 1.5×ULN
* BUN≤ 1.5×ULN
* Signed written informed consent

Exclusion Criteria:

* squamous carcinoma or small cell lung cancer
* Patients were allergic to pemetrexed
* Patients received chemotherapy before
* Uncontrolled acute infection

  .Uncontrolled pleural effusion
* Severe symptomatic heart disease
* Severe infection or metabolic disfunction
* Patients with other malignant tumor
* Uncontrolled brain metastases
* Patients have accepted other clinical trials
* Female patients during their pregnant and lactation period, or patients without contraception

  * Mental disorientation of disorder
  * Glucocorticoids taboo

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
PFS | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhao X, Yu H, Zhao J, Wu X, Sun S, Luo Z, Wang H, Qiao J, Chang J, Wang J. Efficacy and safety of first-line pemetrexed plus carboplatin followed by single-agent pemetrexed maintenance in elderly Chinese patients with non-squamous non-small-cell lung cancer. Oncotarget. 2017 Sep 23;8(49):86384-86394. doi: 10.18632/oncotarget.21186. eCollection 2017 Oct 17. PMID 29156802